CLINICAL TRIAL: NCT00563290
Title: A Phase 2 Study of Dasatinib in Patients With Transplant and Non-Transplant Related Unresectable or Metastatic Cutaneous Squamous Cell Carcinoma and RAI Stage 0-1 Chronic Lymphocytic Leukemia
Brief Title: Dasatinib in Treating Patients With Unresectable or Metastatic Squamous Cell Skin Cancer or RAI Stage 0-I Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00226; NCI-2009-00226 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000576527; OSU-07070; OSU 07070 (Other: Ohio State University Medical Center); 7813 (Other: CTEP); P30CA016058 (NIH); N01CM00070 (NIH)
Record Dates: First submitted 2007-11-22; First posted 2007-11-26 (Estimated); Results first posted 2015-03-20 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-03

CONDITIONS: Recurrent Skin Cancer; Squamous Cell Carcinoma of the Skin; Stage 0 Chronic Lymphocytic Leukemia; Stage I Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Skin Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (dasatinib 100 mg PO BID) (Experimental): Patients receive 100 mg dasatinib PO BID on days 1-28
  Interventions: Drug: dasatinib; Other: laboratory biomarker analysis
- Arm II (dasatinib 70 mg PO BID) (Experimental): Patients receive 70 mg dasatinib PO BID on days 1-28
  Interventions: Drug: dasatinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well dasatinib works in treating patients with unresectable or metastatic squamous cell skin cancer or RAI Stage 0-I chronic lymphocytic leukemia. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate (complete response and partial response) in patients with unresectable or metastatic squamous cell carcinoma of the skin or RAI stage 0-I chronic lymphocytic leukemia receiving dasatinib.

SECONDARY OBJECTIVES:

I. Determine the progression-free survival of patients receiving this drug. II. Evaluate tumor for presence of total EphA2 and both total and active Src and FAK by immunohistochemistry (IHC) pre-treatment with dasatinib.

III. Evaluate tumor for presence of cyclooxygenase-2 by IHC pre-treatment with dasatinib.

OUTLINE: Patients are assigned to 1 of 2 treatment arms.

ARM I: Patients receive 100 mg dasatinib orally (PO) twice daily (BID) on days 1-28.

ARM II (PATIENTS ENROLLED AFTER 11/18/08): Patients receive 70 mg dasatinib PO BID on days 1-28.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Pre-therapy tumor biopsy specimens are collected to detect total and phosphorylated Src and FAK, total EphA2, and cyclooxygenase-2 by immunohistochemistry.

After completion of study treatment, patients are followed up monthly for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following

  * Histologically or cytologically confirmed squamous cell carcinoma of the skin

    * Unresectable or metastatic disease
    * Squamous cell histology represents ≥ 50% of the biopsy specimen
    * May or may not be related to autologous or allogeneic organ transplantation
  * Chronic lymphocytic leukemia (CLL)

    * RAI stage 0-I
    * Stable disease
* Patients with basalosquamous cell disease (basal cell with squamous differentiation) are eligible
* Measurable disease, defined as at least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Must be willing to undergo a pre-treatment tumor biopsy
* Brain metastases are allowed provided the following are true:

  * Received definitive therapy consisting of external beam radiation therapy, gamma knife therapy, or surgical resection resulting in clinically stable disease
  * Lesions are under control for at least 4 weeks after completion of definitive therapy, as measured by repeat MRI or CT scans
  * No requirement for dexamethasone
* ECOG performance status 0-1 OR Karnofsky 60-100%
* Life expectancy > 6 months
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelets ≥ 100,000/mm^3
* Total bilirubin ≤ 1.5 times upper limit of normal(ULN)
* AST/ALT ≤ 2.5 times ULN
* Potassium 3.5 - 5.1 mmol/L
* Calcium > lower limit of normal
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* No known HIV 1 or HIV 2 positivity
* No known hepatitis C or hepatitis B positivity
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to dasatinib
* No QTc prolongation, defined as a QTc interval of ≥ 480 msecs or other significant ECG abnormality
* No condition that impairs the ability to swallow and retain dasatinib tablets (e.g., gastrointestinal tract disease resulting in an inability to take oral medication, requirement for IV alimentation, prior surgical procedure affecting absorption, or active peptic ulcer disease)
* No clinically significant cardiovascular disease including the following:

  * Myocardial infarction within 6 months
  * Uncontrolled angina within 3 months
  * Diagnosed or suspected congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, or Torsades de Pointe)
  * Any history of second or third degree heart block (may be eligible if the subject currently has a pacemaker)
  * Heart rate consistently < 50 beats/minute on pre-entry ECG
  * Uncontrolled hypertension
  * Ejection fraction < 45% by transthoracic echo
* No uncontrolled intercurrent illness including, but not limited to, the following:

  * Ongoing or active infection requiring intravenous antibiotics
  * History of significant bleeding disorder, including congenital (von Willebrand's disease) or acquired (anti-factor VIII antibodies) disorders
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No prior malignancy except for adequately treated basal cell cancer, carcinoma in situ of the cervix, or other cancer for which the patient has been disease free for 3 years
* No gastro-esophageal reflux disease dependent on proton pump inhibitors, H2 blockers, or antacids
* Recovered from prior therapy
* No more than 1 prior therapy with a monoclonal antibody
* No more than 1 prior chemotherapy regimen
* No prior tyrosine kinase inhibitor therapy

  * Prior erlotinib hydrochloride allowed
* More than 2 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) and recovered
* At least 4 weeks since prior radiotherapy

  * Measurable disease must be outside the radiotherapy port
* At least 2 weeks since prior topical therapy
* At least 4 weeks since prior surgery requiring general anesthesia and intubation
* At least 120 days (4 months) since prior amiodarone
* At least 7 days since prior and no concurrent anti-thrombotic and/or platelet agents (e.g., warfarin, heparin, low molecular weight heparin, aspirin [full dose and 81 mg dose] and/or ibuprofen)
* At least 7 days since prior and no concurrent agents with pro-arrhythmic potential
* More than 7 days or 5 half lives, whichever is greater, since prior and no concurrent agents or substances that induce or inhibit CYP3A4
* No concurrent bisphosphonate therapy for the first 8 weeks of dasatinib treatment
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-11; Primary Completion 2012-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Olencki, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I Dasatinib: Patients receive 100 mg orally twice a day.
- Arm II Dasatinib: Patients receive 70 mg dasatinib PO BID on days 1-28
Period: Overall Study
Arm/Group | Arm I Dasatinib | Arm II Dasatinib
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I Dasatinib: Patients receive oral dasatinib 100 mg twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm II Dastinib: Patients receive oral dasatinib 70 mg twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Arm I Dasatinib | Arm II Dastinib | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 5
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Complete Response and Partial Response)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Every 2 courses during treatment, assessed up to 12 weeks after completion of treatment
Measure: Number; unit: percentage of patients
Groups:
- Arm I: Dasatinib: Patients receive 100 mg orally twice a day.
- Arm II: Dasatinib: Patients receive 70 mg orally twice a day.
Arm/Group | Arm I: Dasatinib | Arm II: Dasatinib
Number analyzed (Participants) | 3 | 4
percentage of patients | 0 | 0

2. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Time from start of treatment to time of progression, assessed up to 12 weeks
Population: The second treatment arm of Dasatinib 70 mg orally twice a day was created as a result of an amendment to the protocol therefore the patient PFS data was combined for each arm.
Measure: Median (Full Range); unit: weeks
Groups:
- Arm I and Arm II: For Arm I patients receive Dasatinib100 mg orally twice a day.
  For Arm II patients receive Dasatinib 70 mg orally twice a day.
Arm/Group | Arm I and Arm II
Number analyzed (Participants) | 7
weeks | 4 [4 to 8]

3. Secondary Outcome: Presence of Total EphA2 and Both Total and Active Src and FAK by Immunohistochemistry (IHC)
Description: Performed per standard protocols by the Pathology Department.
Time Frame: At baseline
Population: Funding was not available to do correlative studies
Groups:
- Dasatinib: Patients receive 100 mg orally twice a day. Due to a dosing update the dose was decreased to 70 mg orally twice a day.
Arm/Group | Dasatinib
Number analyzed (Participants) | 0

4. Secondary Outcome: COX-2 Presence by IHC
Description: Performed per standard protocols by the Pathology Department. Samples will be obtained pre-therapy. Determination of the COX-2 tumor status on this trial will develop the beginnings of a data base upon which future therapy may be designed.
Time Frame: At baseline
Population: Funding was not available to do correlative studies
Arm/Group | Dasatinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Patients will be evaluated for Adverse Events from week 1 up until 12 weeks.
Description: Toxicities were graded using the Common Toxicity Criteria Version 3.0 (CTC 3.0)
Groups:
- Dasatinib 100 mg: Patients receive the initial dose of 100 mg orally twice a day.
- Dasatinib 70 mg: Patients receive the initial dose of 70 mg orally twice a day. Dose was reduced to 70 mg orally based on toxicity.
Arm/Group | Dasatinib 100 mg | Dasatinib 70 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 1/3 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib 100 mg (N=3) | Dasatinib 70 mg (N=4)
Hemorrhage/Bleeding (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0)
Vascular- other (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — unknown ANC
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) — unknown ANC

LIMITATIONS AND CAVEATS:
3 patients were treated with Dasatinib 100 mg PO twice daily and 4 patients were treated with Daatinib 70 mg PO twice daily.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less